CLINICAL TRIAL: NCT05245994
Title: An Open Label, Multicenter Phase 2 Study of Durvalumab (MEDI4736) + Olaparib as Maintenance Therapy in Patients With Extensive Stage Small-Cell Lung Cancer
Brief Title: An Open Label, Multicenter Phase 2 Study of Durvalumab (MEDI4736) + Olaparib as Maintenance Therapy in Chinese
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Zhang, MD (Other)
Responsible Party: Sponsor-Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-20-20659
Record Dates: First submitted 2022-01-23; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer; Small Cell Lung Cancer; Durvalumab
Keywords: ES-SCLC; Durvalumab; Olaparib
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — durvalumab; Etoposide; Cisplatin; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab, etoposide, and cisplatin/carboplatin followed by durvalumab and olaparib (Experimental)
  Interventions: Drug: Durvalumab, etoposide, and cisplatin/carboplatin followed by durvalumab and olaparib

INTERVENTIONS:
Drug: Durvalumab, etoposide, and cisplatin/carboplatin followed by durvalumab and olaparib — Durvalumab 1500 mg intravenous infusion, started to be used simultaneously with chemotherapy at week 0 and continued after chemotherapy. Starting from week 0, the dose of etoposide + carboplatin or cisplatin in the study will not exceed the dose for specific indications in the product instructions (etoposide [80 to 100mg/m2] via intravenous infusion and carboplatin [ The area under the curve (AUC) is 5-6] by intravenous infusion or cisplatin [75-80 mg/m2] by intravenous infusion), using up to 4 cycles. The choice of platinum drugs is at the discretion of the investigator. The initial dose of olaparib is 300mg twice daily. Olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water. The tablets should be swallowed whole and not chewed, crushed, dissolved or divided. Olaparib tablets can be taken with or without food.

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of combining durvalumab with EP followed by durvalumab + olaparib maintenance therapy as first-line treatment in patients with extensive-disease small-cell lung cancer (SCLC).

DETAILED DESCRIPTION:
This study is planned to enroll approximately 60 eligible patients in China. Patients who fulfill all the inclusion criteria and none of the exclusion criteria will receive 4 cycles of EP with durvalumab, then durvalumab + olaparib will be administered post-chemotherapy until confirmed progressive disease (PD).Tumor assessments will be performed at Screening as baseline with follow-up at Week 6 ±1 week from the date of the first cycle treatment, at Week 12 ±1 week from the date of the first cycle treatment, and then every 8 weeks ±1 week until confirmed objective disease progression. The primary endpoint is APF12, which is defined as the Proportion of patients alive and progression free at 12 months from the first date of the first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years at the time of screening.
2. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
3. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
4. Histologically or cytologically documented extensive disease (American Joint Committee on Cancer Stage (7th edition) IV SCLC [T any, N any, M1 a/b]), or T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan.

   Brain metastases; must be asymptomatic or treated and stable off steroids and anti-convulsants for at least 1 month prior to study treatment. Patients with suspected brain metastases at screening should have a CT/MRI of the brain prior to study entry.
5. Provision of an archived tumor tissue block (or at least 15 newly cut unstained slides) where such samples exist.
6. Patients must be considered suitable to receive a platinum based chemotherapy regimen as 1st line treatment for the ED-SCLC. Chemotherapy must contain either cisplatin or carboplatin in combination with etoposide.
7. Life expectancy ≥16 weeks at Day 1.
8. World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2 at enrollment. PS2 patients are permitted to receive first-line treatment, and PS score should be reassessed after first-line treatment. Then patients who are assessed as PS2 at the completion of chemotherapy+durvalumab will be excluded.
9. Body weight >30 kg.
10. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have a short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines.
11. No prior exposure to immune-mediated therapy including, but not limited to, other PARP inhibitor, anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.
12. Adequate organ and marrow function which is measured within 28 days prior to administration of study treatment as defined below:

    Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days Absolute neutrophil count ≥1.5 × 109/L (use of granulocyte colony-stimulating factor is not permitted at screening).

    Platelet count ≥100 × 109/L. Serum bilirubin ≤1.5 × the upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physicians.

    In patients without hepatic metastasis: ALT and AST ≤2.5 × ULN. In patients with hepatic metastases, ALT and AST ≤5 × ULN.

    Measured or calculated creatinine clearance: >60mL/min for patients on cisplatin and >51mL/min for patients on carboplatin, as determined by Cockcroft-Gault (using actual body weight) or based on a 24 hour urine test:

    Males:

    Creatinine CL (mL/min) = [Weight (kg) × (140 - Age)] / [72 × Serum creatinine (mg/dL)]

    Females:

    Creatinine CL (mL/min) = {[Weight (kg) × (140 - Age)] / [72 × Serum creatinine (mg/dL)]}*0.85
13. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    Women <50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

    Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
14. Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception

Exclusion Criteria:

1. Previous IP assignment in the present study.
2. Concurrent enrollment in another clinical study, unless it is an observational (non interventional) clinical study or during the follow up period of an interventional study.
3. Participation in another clinical study with an IP during the last 4 weeks.
4. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
5. Medical contraindication to etoposide platinum (carboplatin or cisplatin) based chemotherapy.
6. Any history of radiotherapy to the chest prior to systemic therapy or planned consolidation chest radiation therapy. Radiation therapy outside of the chest for palliative care (ie, bone metastasis) is allowed but must be completed before first dose of the study medication.
7. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (eg, hormone replacement therapy) is acceptable.
8. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
9. History of allogeneic organ transplantation.
10. Has a paraneoplastic syndrome (PNS) of autoimmune nature, requiring systemic treatment (systemic steroids or immunosuppressive agents) or has a clinical symptomatology suggesting worsening of PNS.
11. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis with the exception of diverticulosis, systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, and uveitis, etc]). The following are exceptions to this criterion:

    Patients with vitiligo or alopecia Patients with hypothyroidism (eg, following Hashimoto syndrome) and stable on hormone replacement Any chronic skin condition that does not require systemic therapy Patients without active disease in the last 5 years may be included but only after consultation with the investigator Patients with celiac disease controlled by diet alone
12. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, interstitial lung disease, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
13. History of another primary malignancy except for Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease Adequately treated carcinoma in situ without evidence of disease
14. History of leptomeningeal carcinomatosis.
15. History of active primary immunodeficiency.
16. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive HBV surface antigen [HbsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or olaparib. The following are exceptions to this criterion:

    Intranasal, inhaled, topical steroids or local steroid injections (eg, intra articular injection).

    Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.

    Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication). Premedication with steroids for chemotherapy is acceptable.
18. Receipt of live, attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
19. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from Screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + olaparib combination therapy.
20. Known allergy or hypersensitivity to durvalumab, olaparib, etoposide, carboplatin, cisplatin, or any of their excipients
21. Prior randomization or treatment in a previous durvalumab and/or olaparib clinical study regardless of treatment arm assignment.
22. *Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.

23. *Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.

24) *Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.

25) *Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.

26) *Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.

27) *Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting Olaprrib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.

28) *Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).

29) *Breast feeding women. 30) Patients with a known hypersensitivity to the combination/comparator agent. 31) As judged by the investigator, any evidence of which in the investigator's opinion makes it undesirable for the patient to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
APF12-Alive and Progression Free | 1 year
  A proportion of patients alive and progression free at 12 months from the first date of first-line treatment

SECONDARY OUTCOMES:
PFS0-Progression Free Survival 0 | 2 years
  The time from the first date of first-line treatment until the date of objective disease progression or death.
PFS-Progression Free Survival | 2 years
  The time from the first date of maintenance treatment until the date of objective disease progression or death.
OS-Overall Survival | 2 years
  The time from the start of first-line treatment to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off.
ORR-Objective Response Rate | 2 years
  Objective response rate after the given treatment in patients accoeding to the evaluation criteria of RECIST1.1.
  Objective response rate after the given treatment according to the evaluation criteria of RECIST1.1

OTHER OUTCOMES:
AE-Adverse Events | 2 years
  Any undesirable medical conditions (other than progression of the malignancy under evaluation) or the deterioration of a pre existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No